CLINICAL TRIAL: NCT03689101
Title: To Explore the Relationship Between Endometrial CD138 Count and Pregnancy Outcome Following Frozen Embryo Transfer in Natural Cycles
Brief Title: The Relationship Between CD138 Count of Endometrium and Reproductive Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P2018009
Record Dates: First submitted 2018-09-21; First posted 2018-09-28 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endometrial biopsies (Experimental): Endometrial biopsy was performed precisely 7 days after LH surge (LH+7) to count endometrial CD138.
  Interventions: Procedure: Endometrial biopsies

INTERVENTIONS:
Procedure: Endometrial biopsies — Endometrial biopsy was performed precisely 7 days after LH surge (LH+7)

SUMMARY:
It's well known, endometritis affects reproductive outcomes. Though CD138 counting as one new diagnosis measure for endometritis, diagnostic criterion of this measure isn't consistent. And if the CD138 counting is correlation to the outcome of reproductive is not clear.

Firstly, This study aims to explore the relationship between endometrial CD138 count and pregnancy outcome following frozen embryo transfer in natural cycles. Secondly , the investigators want to find a cut-off value which is related to reproduction outcome.

ELIGIBILITY:
Inclusion Criteria:

* age between20 and 38 years;
* regular menstrual cycles;
* body mass index (BMI) ranged from 18 to 25

Exclusion Criteria:

* uterine abnormalities;
* intrauterine adhesions（moderate - severe）, advanced endometriosis, adenomyosis, untreated hydrosalpinx, uterine fibroids (submucosal fibroids, nonmucosal fibroids >4.0 cm and/or endometrial pressure)

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
CD138 counting | 7 days after LH surge (LH+7)
clinical pregnancy rate | about 28 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Fei Gong, doctor, Principal Investigator — Reproductive & Genetic Hospital of CITIC-Xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China